CLINICAL TRIAL: NCT03909243
Title: Assessment of Child Psychological Attributes Using Strength and Difficulties Questionnaire for Prediction of Child Behavior at First Dental Visit Through: A Cross Sectional Study
Brief Title: Assessment of Child Psychological Attributes for Prediction of Child Behavior at First Dental Visit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandra Moussa Anwar, Principal investigator, Cairo University
Other Study IDs: 14422017495365
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Psychological Disorders
Keywords: psychological attributes; child mental disorders; strength and difficulties questionnaire; child behavior
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders; Child Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One of the most prevalent chronic diseases worldwide is mental disorder, including social, emotional, and behavioral problems, and it is the fifth main cause of global disability . In Egypt, it is estimated that 20.6% of children aged from 6-12 years had behavioral problems

Behavioral and emotional problems may affect deeply child's quality of life, such as impairment of school life (high absence), They may cause nutritional imbalance and even suicidal thoughts. Therefore, both the dentist and the family should be adequately prepared to deal with those children who come seeking dental treatment.

Recently, studies proved the association between the psychological characteristics and the behavior of children in dental setting. There was a study that showed that there is a relation between psychological functioning of the child, dental anxiety and his/her behaviour during dental appointment. Furthermore, it was found that there is a correlation between the temperamental difficulties or emotional problems of the child and the non-cooperative behavior during the process of injection of the local anesethia.

These studies ensures the importance of understanding the effect of mental disorders on the behavior of children during dental treatment, as it would help the professionals to properly plan the clinic appointments without any delay or cancellation of the appointment and allows him to render effective and efficient dental treatment.

DETAILED DESCRIPTION:
this study aims to acknowledge the different psychological attributes among children seeking dental treatment at young age and to assess the association between child psychological attributes and his/her behavior in dental clinic.

ELIGIBILITY:
Inclusion Criteria:

* Children: school aged children (4 to 7) years old
* Teeth: carious teeth requiring a simple dental treatment (cavity preparation with restoration)

Exclusion Criteria:

* Children:

  * Medically compromised children.
  * Children with previous dental history.
  * Refusal of participation.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Out patients of Pediatric Dentistry and Dental Public Health Department at Faculty of Dentistry, Cairo University, Egypt who are having a dental problem and coming for their first dental visit.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Child psychological attributes | 6 months
  Total difficulty score using strengths and difficulties questionnaire (0-40)
  0-13 normal
  14-16 border line
  17-40 abnormal

SECONDARY OUTCOMES:
Actual child behavior during the dental treatment. | 6 months
  Rating (0-4) using Fankl scale
  Rating 1 (--) definitely negative Refusal of treatment, forceful crying, fearfulness or any other overt evidence of extreme negativism.
  Rating 2 (-) negative Reluctance to accept treatment, uncooperativeness, some evidence of negative attitude but not pronounced.
  Rating 3 (+) positive Acceptance of treatment, cautious behaviour at times willingness to comly with the dentist, at times with reservation, but patient follows the dentist's directions cooperatively.
  Rating 4 (++) definitely positive Good rapport with the dentist, interest in the dental procedure, laughing and enjoying the situation.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Anwar, BSc, Principal Investigator — Resident at pediatric Dentistry and Dental Public Health Department; Sara A Mahmoud, phD, Study Director — Associate professor at pediatric Dentistry and Dental Public Health Department